CLINICAL TRIAL: NCT04610294
Title: Operating Room Air Filtration/Sterilization and Surgical Site Infection: A Randomized Multiple Cross-over Cluster Trial
Brief Title: Operating Room Air Filtration/Sterilization
Acronym: ORACLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20-656
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Surgery
MeSH Terms: interventions — Sterilization, Reproductive

STUDY DESIGN:
Intervention Model Description: Randomized multiple crossover cluster trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical-looking test devices are either active or inactive. None of the investigators, clinicians, patients, or outcome assessors knows which are which.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Aerus air sterilization (Experimental): Aerus air sterilization system will be used in an operating room, in addition to routine room air filtration
  Interventions: Device: Functioning Aerus air filtration/sterilization
- Conventional air handling (Active Comparator): Only routine room air filtration will be used in an operation room.
  Interventions: Device: Deactivated Aerus air filtration/sterilization

INTERVENTIONS:
Device: Functioning Aerus air filtration/sterilization — Two units of Aerus air sterilization system will be used in each operating room, and each will be set to "high." Units used for the trial will be modified internally to be active and will be sealed to prevent operating room personnel from opening the system and determining a unit's status.
  Arms: Aerus air sterilization
Device: Deactivated Aerus air filtration/sterilization — Two units of Aerus air sterilization system will be used in each operating room, and each will be set to "high." Units used for the trial will be modified internally to be inactivated and will be sealed to prevent operating room personnel from opening the system and determining a unit's status. Units will be inactivated by removing the activated carbon, high-efficiency particulate filter, and ionization chamber. However, the fan will remain active as will the "run" lights.
  Arms: Conventional air handling

SUMMARY:
Determine whether operating room air filtration and sterilization with the ActivePure system reduces a composite of serious surgical site infections, infection-related complications, and death within 30 days after surgery.

DETAILED DESCRIPTION:
The investigators primary goal is thus to determine whether supplemental filtering and sterilizing operating room air reduces a composite of serious surgical site infections, infection-related complications, and death within 30 days after surgery. The primary outcome will be restricted to inpatients. However, outpatients will be simultaneously enrolled given the trial's cluster design. Sample-size is based on our primary inpatient analysis, N= 66,273 inpatients. Available outpatients will be included for analysis of our secondary outcome which includes both inpatients and outpatients.

ELIGIBILITY:
Inclusion Criteria:

* All patients in designated adult operating rooms
* American Society of Anesthesiologists physical status 1-4.
* Surgery lasting at least 1 hour.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66273 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Serious surgical site infections and related complication in previously uninfected surgical inpatients | 30 days after surgery
  Composite of serious surgical site infections, infection-related complications, and death in surgical inpatients without present-on-admission composite infection components

SECONDARY OUTCOMES:
Serious surgical site infections and related complication in previously uninfected surgical inpatients and outpatients | 30 days after surgery
  Composite of serious surgical site infections, infection-related complications, and death in surgical inpatients and outpatients without present-on-admission composite infection components

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient level data will be shared collaboratively. Sharing will require approval of the trial steering committee and appropriate institutions approvals and data-sharing contracts.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 1 year after publication of the main trial paper.
Access Criteria: Contact principal investigator.